CLINICAL TRIAL: NCT02701738
Title: Impact of Exercise on the Metabolic Consequences of Overeating
Acronym: XO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Professor, Movement Science and Director, Substrate Metabolism Laboratory, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00102772
Record Dates: First submitted 2016-01-21; First posted 2016-03-08 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overeating Protocol (Experimental): Subjects will ingest 30% more calories per day than their calculated daily energy requirements (~750kcals extra energy intake each day). All subjects will be instructed (and will be guided) to consume a diet containing approximately 50% carbohydrate, 35% fat, and 15% protein.
  Interventions: Dietary Supplement: Overeating Protocol

INTERVENTIONS:
Dietary Supplement: Overeating Protocol — Subjects will ingest 30% more calories per day than their calculated daily energy requirements (~750kcals extra energy intake each day). All subjects will be instructed (and will be guided) to consume a diet containing approximately 50% carbohydrate, 35% fat, and 15% protein.

SUMMARY:
The primary purpose of this study is to examine the effects of 1-week of overeating on important clinical metabolic health outcomes (e.g., glucose tolerance, blood lipid profile, and blood pressure) and factors regulating the structure and metabolic function of fat tissue. This study will determine how regular exercise during this overeating period impacts these responses.

DETAILED DESCRIPTION:
If subjects are eligible and decide to participate, they will take part in two identical study trials. One is scheduled before and the other is scheduled after 1 week of overeating controlled by the study team. Subjects who exercise regularly will be instructed to exercise the day before their first study trial - and they will be required to exercise during 6 of the 7 days of the overeating period (including the day before their second study trial). Subjects who do not regularly exercise (no planned physical activity) will remain inactive until the completion of both study trials.

Before each study trial If a subject is a regular exerciser, they will be asked to come to the Substrate Metabolism Laboratory in the afternoon before each of the 2 study trials to exercise in the lab for 45 min at a moderate intensity. The evening before the study trial, all subjects will need to eat a standardized dinner meal and snack. They must eat the meal and snack at specific times as indicated by the research staff. After eating the snack, subjects will need to fast (no food or beverages - besides water) overnight.

During each study trial Subjects will arrive at the Substrate Metabolism Laboratory at 7:00AM and will rest quietly for approximately 30 min. After which, the study team will measure their resting blood pressure and their resting metabolic rate. An intravenous catheter (IV) will then be placed in a vein of the subject's hand or forearm for blood sampling. The research team will then collect a small sample of fat tissue in the subject's abdomen with a needle. Next, subjects will drink a sweet sugar solution for an Oral Glucose Tolerance Test (OGTT) and the research team will collect blood samples every 15 min for 3 hours. After this 3 hour test, the IV catheter will be removed and subjects will be provided breakfast and discharged.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40
* Body Mass Index: 20-30 kg/m2
* Exercise group: (≥5 days/wk of aerobic exercise; 30-60min/session at moderate and vigorous intensities)
* No Exercise group: no regularly planned exercise/physical activity
* Women must have regularly occurring menses and must be premenopausal

Exclusion Criteria:

* Pregnant or lactating
* Blood pressure > 140/90 mm Hg
* Evidence/history of cardiovascular or metabolic disease
* Medications known to affect lipid or glucose metabolism
* Tobacco or electronic cigarette user

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01-12; Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Oral Glucose Tolerance | up to 1 week
  An index of insulin sensitivity will be measured using the plasma insulin and glucose concentrations during the 3h OGTT

SECONDARY OUTCOMES:
Resting Metabolic Rate | baseline and 1 week
Total Cholesterol | baseline and 1 week
  Plasma concentrations of total- cholesterol will be measured
PPARg mRNA expression | baseline and 1 week
  cytokine proteins will be measured in adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Ludzki AC, Krueger EM, Gillen JB, Taylor NM, Middlebrook DO, Baldwin TC, Karabetsos KC, Schleh MW, Horowitz JF. One week of overeating upregulates angiogenic and lipolytic gene expression in human subcutaneous adipose tissue from exercise trained and untrained adults. Appl Physiol Nutr Metab. 2022 Oct 1;47(10):992-1004. doi: 10.1139/apnm-2022-0078. Epub 2022 Jul 11. PMID 35816737